CLINICAL TRIAL: NCT02294019
Title: A Multicenter Actual Use And Compliance Study Of Ibuprofen 400 Mg In A Simulated Over-the-counter Environment
Brief Title: Actual Use Trial of Ibuprofen 400 mg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None
Other Study IDs: B3491013; AUT (Other: Alias Study Number)
Record Dates: First submitted 2014-11-14; First posted 2014-11-19 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-04

CONDITIONS: Patient Compliance
Keywords: ibuprofen 400 mg; actual use; compliance
MeSH Terms: conditions — Patient Compliance | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ibuprofen caplet arm (Experimental)
  Interventions: Drug: Ibuprofen 400 mg caplet

INTERVENTIONS:
Drug: Ibuprofen 400 mg caplet — 400 milligram (mg) caplet according to Drug Facts label

SUMMARY:
This is an open label, multicenter, 30 day study designed to mimic an OTC like environment in which subjects will use the product after making a purchase decision about ibuprofen 400 mg caplets based only on their reading of the Drug Facts Label (DFL) and other information on the package.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age (19 years of age in Alabama)
* Subject reports taking over-the-counter (OTC) analgesics for pain or fever relief

Exclusion Criteria:

* Current government-issued identification (ID)
* Pregnant or breastfeeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 738 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- United States (25):
  - Robert's Discount Pharmacy, Hoover, Alabama
  - Pharmacy at the Pig, McCalla, Alabama
  - Community Clinical Pharmacy, Mesa, Arizona
  - Garden Drug, Fort Lauderdale, Florida
  - Pill Box Pharmacy and Medical Supply, Pembroke Pines, Florida
  - Summerfield Pharmacy, Riverview, Florida
  - Sutton Family Pharmacy, Dalton, Georgia
  - Wynn's Pharmacy Inc., Griffin, Georgia
  - Goodrich Pharmacy, Andover, Minnesota
  - Goodrich Pharmacy, Anoka, Minnesota
  - Goodrich Pharmacy, Blaine, Minnesota
  - Goodrich Pharmacy, Elk River, Minnesota
  - Cub Pharmacy Number 1924, Saint Louis Park, Minnesota
  - Albers' Specialty Pharmacy, Kansas City, Missouri
  - Countryside Pharmacy, Savannah, Missouri
  - Texas Road Pharmacy, Monroe, New Jersey
  - Phil's Pills, Inc., Albuquerque, New Mexico
  - Total Health and Wellness Center of Taos, Taos, New Mexico
  - Kroger Pharmacy #342, Cary, North Carolina
  - Family Prescription Center, Bethlehem, Pennsylvania
  - The Medicine Shoppe, Bountiful, Utah
  - Northview Pharmacy, Layton, Utah
  - Family Plaza Pharmacy, West Jordan, Utah
  - Foothills Compounding Pharmacy, Enumclaw, Washington
  - Ostrom Drugs, Kenmore, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3491013&StudyName=A%20Multicenter%20Actual%20Use%20And%20Compliance%20Study%20Of%0Aibuprofen%20400%20Mg%20In%20A%20Simulated%20Over-the-counter%20Environment

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were screened by phone,then referred to their participating retail pharmacy site for scheduled face-to-face interview,after which they were given an empty ibuprofen 400 milligram (mg) caplet over-the-counter (OTC) package to review information on outside of entire package,then decision was made to purchase medicine by them.
Groups:
- Ibuprofen: All participants who purchased at least 1 carton of study medication.
Period: Overall Study
Arm/Group | Ibuprofen
Started | 738
Completed | 635
Not Completed | 103
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 68
Not completed — Lost to Follow-up | 31
Not completed — Other | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All participants who purchased at least 1 carton of study medication.
Arm/Group | Ibuprofen
Number analyzed (Participants) | 738
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 412
  Male | 326

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Taking Greater Than (>) 1200 Milligram (mg) (>3 Caplets) on no More Than 2 Use Days During the Study
Description: Percentage of participants whose behavior was either correct or acceptable were considered to be compliant. The behavior was considered correct if participants took more than 1200 mg (>3 caplets) on either 0, 1 or 2 use days (where a use day was defined as a calendar day starting at 12:01 AM in which a participant received at least one dose of study medication), based on their diary. The behavior was considered acceptable if a participant exceeded the labelled daily dosing directions of taking more than 3 caplets per day, under the advice of a healthcare professional, based on information from the end of study follow-up interview.
Time Frame: Day 1 up to 30 days
Population: Actual use population included all participants who purchased the study medication and recorded the use of study medication in the diary on or after the first purchase date, and returned the diary.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Ibuprofen: Participants who purchased and used orally 400 mg caplets of Ibuprofen after reading the drug facts label (DFL), and recorded the use of study medication in the diary on or after the first purchase date, and returned the diary.
Arm/Group | Ibuprofen
Number analyzed (Participants) | 685
percentage of participants | 95.2 [93.6 to 96.8]

2. Secondary Outcome: Percentage of Participants Taking Greater Than (>) 400 mg (>1 Caplet) at a Time on no More Than 2 Dosing Occasions During the Study
Description: Percentage of participants whose behavior was either correct or acceptable were considered to be compliant. The behavior was considered correct if the total number of dosing occasions (distinct usage date/time values from their diary) in which a participant received 2 or more caplets was 0, 1 or 2. The behavior was considered acceptable if a participant exceeded the labelled daily dosing directions of taking no more than 1 caplet per dose, under the advice of a healthcare professional, based on the end of study follow up interview.
Time Frame: Day1 up to 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ibuprofen
Number analyzed (Participants) | 685
percentage of participants | 84.4 [81.7 to 87.1]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant or one participant may have experienced both a serious and non-serious event during the study.
Groups:
- Ibuprofen (Safety Population): Subjects in the actual use population, and any other subject who provided any follow up information indicating that they used the study product at least once during the study
Arm/Group | Ibuprofen (Safety Population)
Serious Adverse Events (participants affected / at risk) | 6/736
Other Adverse Events (participants affected / at risk) | 76/736
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibuprofen (Safety Population) (N=736)
Coronary artery occlusion (Cardiac disorders) | 1
Atypical pneumonia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibuprofen (Safety Population) (N=736)
Palpitations (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Eye irritation (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Haematochezia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Pancreatitis acute (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 2
Peripheral swelling (General disorders) | 1
Atypical pneumonia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Influenza (Infections and infestations) | 3
Localised infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 8
Pharyngitis streptococcal (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 1
Sialoadenitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Wound infection (Infections and infestations) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Eye injury (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 3
Ligament sprain (Injury, poisoning and procedural complications) | 2
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Blood pressure increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 3
Migraine (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Anger (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Libido decreased (Psychiatric disorders) | 1
Renal pain (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.